CLINICAL TRIAL: NCT02735421
Title: Effect of Adapalene 0.3% - Benzoyl Peroxide 2.5% Gel Versus Vehicle Gel on the Risk of Formation of Atrophic Acne Scars in Moderate to Severe Acne Subjects
Brief Title: Adapalene 0.3% - Benzoyl Peroxide 2.5% Gel and Risk of Formation of Atrophic Acne Scars
Acronym: OSCAR
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Galderma R&D (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: RD.03.SPR.105061; 2016-002666-31 (EudraCT Number)
Record Dates: First submitted 2016-04-07; First posted 2016-04-12 (Estimated); Results first posted 2019-11-15 (Actual); Last update posted 2022-09-14 (Actual); Status verified 2022-08

CONDITIONS: Acne Vulgaris; Atrophic Acne Scars
Keywords: acne; scars
MeSH Terms: conditions — Acne Vulgaris; Cicatrix

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Part 1: ABPO Forte Gel (Experimental)
  Interventions: Drug: ABPO Forte Gel
- Part 1: ABPO Forte Vehicle Gel (Placebo Comparator)
  Interventions: Drug: Vehicle gel
- Part 2: ABPO Forte Gel (Experimental)
  Interventions: Drug: ABPO Forte Gel
- Part 2: ABPO Forte Vehicle Gel (Placebo Comparator)
  Interventions: Drug: Vehicle gel

INTERVENTIONS:
Drug: ABPO Forte Gel — Participants applied Adapalene 0.3% - Benzoyl peroxide (BPO) 2.5% gel (ABPO Forte) topically to the affected areas once daily for 24 weeks in Part 1 and for 48 weeks in Part 2.
  Other Names: TactuPump Forte
  Arms: Part 1: ABPO Forte Gel; Part 2: ABPO Forte Gel
Drug: Vehicle gel — Participants applied placebo matched to ABPO Forte gel topically to the affected areas once daily for 24 weeks in Part 1 and 48 weeks in Part 2.
  Arms: Part 1: ABPO Forte Vehicle Gel; Part 2: ABPO Forte Vehicle Gel

SUMMARY:
This was a multi-centre, randomized, investigator blinded, vehicle controlled trial using intra-individual comparison (right half-face versus left half-face).

Participants with each half-face randomized to one of the two following treatments:

* Adapalene 0.3 percent (%) - benzoyl peroxide (BPO) 2.5% gel (TactuPump® Forte).
* Vehicle gel

The main objective of this trial was to evaluate the effect of Adapalene 0.3% - BPO 2.5% (ABPO Forte) gel versus vehicle gel on the risk of formation of atrophic acne scars in moderate to severe acne participants.

ELIGIBILITY:
Main Inclusion Criteria:

* Participants with clinical diagnosis of moderate to severe acne vulgaris on the face defined by:

  1. Investigator's Global Assessment score of 3 or 4, with same score on both sides; and
  2. A minimum of 25 inflammatory lesions (papules and pustules) in total, with at least 10 on each side (excluding the nose); and
  3. No more than two acne nodules (less than or equal to [>=] 1 centimeter [cm]); and
  4. A minimum of 10 atrophic acne scars in total (upper than 2 millimeters [mm]) (excluding the nose)
* Participants with a symmetric number of both inflammatory and non-inflammatory lesions on the whole face, and atrophic acne scars on the whole face.
* Participants with skin phototype of I to IV on Fitzpatrick's scale.

Main Exclusion Criteria:

* Participants with acne conglobata, acne fulminans, secondary acne (chloracne, drug-induced acne, etc.), nodulo cystic acne, acne requiring systemic treatment.
* Prior failure to treatment with TactuPump® Forte (Adapalene 0.3% - BPO 2.5%).
* Participants with more than 3 excoriated acne lesions.
* Participants with skin abraded on the treated area or affected by eczema, seborrhoeic dermatitis, cuts or sunburn.
* Female participant who is pregnant, nursing or planning a pregnancy during the trial or within one month after the last trial treatment application.
* Male participant with a beard or facial hair, which would interfere with the clinical trial evaluations or clinical trial procedures.
* Participants having received at least one of the following topical treatments on the treated area: Corticosteroids, antibiotics, benzoyl peroxide, azelaic acid, hydroxyacids, Zinc containing treatments, antibacterials, antiseptics, other anti-inflammatory drugs or other acne treatments (2 weeks); Retinoids (4 weeks); Cosmetic/aesthetic procedures on the face (1 week); Photodynamic therapy, laser therapy, microdermabrasion for acne (3 months).
* Participants having received at least one of the following systemic treatments: Corticosteroids (except locally acting corticosteroids such as inhaled or intrathecal or dermal application at distance from the face), antibiotics (except penicillin) (1 month); Spironolactone (3 months) / Drospirenone (3 months, unless dose is stable since at least 3 months); Oral retinoids (6 months); Cyproterone acetate / Chlormadinone acetate (6 months); Immunomodulators (3 months).

Ages: 16 Years to 35 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 67 (Actual)
Dates: Start 2016-05-13 (Actual); Primary Completion 2017-06-05 (Actual); Study Completion 2017-11-23 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- Canada (6):
  - Markham, Ontario
  - Oakville, Ontario
  - Toronto, Ontario
  - Windsor, Ontario
  - Montreal, Quebec
  - Saint-Jérôme, Quebec
- Nantes, France

REFERENCES:
- [Background] Dreno B, Bissonnette R, Gagne-Henley A, Barankin B, Lynde C, Chavda R, Kerrouche N, Tan J. Long-Term Effectiveness and Safety of Up to 48 Weeks' Treatment with Topical Adapalene 0.3%/Benzoyl Peroxide 2.5% Gel in the Prevention and Reduction of Atrophic Acne Scars in Moderate and Severe Facial Acne. Am J Clin Dermatol. 2019 Oct;20(5):725-732. doi: 10.1007/s40257-019-00454-6. PMID 31209851
- [Background] Dreno B, Bissonnette R, Gagne-Henley A, Barankin B, Lynde C, Kerrouche N, Tan J. Prevention and Reduction of Atrophic Acne Scars with Adapalene 0.3%/Benzoyl Peroxide 2.5% Gel in Subjects with Moderate or Severe Facial Acne: Results of a 6-Month Randomized, Vehicle-Controlled Trial Using Intra-Individual Comparison. Am J Clin Dermatol. 2018 Apr;19(2):275-286. doi: 10.1007/s40257-018-0352-y. PMID 29549588

RESULTS

PARTICIPANT FLOW:
Recruitment Details: The study was conducted at 6 centers in Canada and France between 13 May 2016 and 23 November 2017. This study was conducted in 2 parts: Part 1 (Randomized) and Part 2 (Open Label).
Pre-assignment Details: A total of 67 participants were randomized. All eligible participants had each half-face randomized to one of the two following treatments (with the other treatment applied to the other side of the face): ABPO forte gel and ABPO forte vehicle gel.
Groups:
- All Participants: Participants applied once-daily adapalene 0.3% - benzoyl peroxide (BPO) 2.5% (ABPO Forte) gel on half-face and ABPO Forte vehicle gel on the other side of the face based on randomization (right or left side of the face) at night for 24 weeks were enrolled in Part 1 of the study. Thereafter, at the decision of the investigator, based on participant's medical assessment of efficacy during Part I, the participants who agreed to continue treatment with ABPO Forte gel for up to 24 additional weeks on the whole face were enrolled in Part 2 of the study.
Period: Part A (Randomized): up to 24 Weeks
Arm/Group | All Participants
Started | 67
Completed | 54
Not Completed | 13
Not completed — Adverse Event | 2
Not completed — Withdrawal by Subject | 6
Not completed — Lost to Follow-up | 3
Not completed — Inadequate compliance to treatment | 1
Not completed — Pregnancy | 1
Period: Part 2 (Open Label): up to 48 Weeks
Arm/Group | All Participants
Started | 45 (Participants who continue treatment with A-BPO Forte gel for up to 24 additional weeks.)
Completed | 41
Not Completed | 4
Not completed — Withdrawal by Subject | 1
Not completed — Lost to Follow-up | 3

BASELINE CHARACTERISTICS:
Population: Intent-to-Treat (ITT) Population included all entire population enrolled and randomized.
Arm/Group | All Participants
Number analyzed (Participants) | 67
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 19
  Between 18 and 65 years | 48
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 21.5 (4.2)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 44
  Male | 23
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0
  Asian | 9
  Native Hawaiian or Other Pacific Islander | 0
  Black or African American | 0
  White | 58
  More than one race | 0
  Unknown or Not Reported | 0
Region of Enrollment [Count of Participants; unit: Participants]
  Canada | 48
  France | 19
Skin Phototype [Count of Participants; unit: Participants] — Fitzpatrick skin phototype is a system used to describe a person's skin type. It ranges from skin phototype I to VI. Where, skin phototype I = pale white skin, blue/green eyes, blond/red hair, always burns, does not tan; skin phototype II = fair skin, blue eyes; burns easily, tans poorly; skin phototype III = darker white skin, tans after initial burn; skin phototype IV = light brown skin, burns minimally, tans easily; skin phototype V = brown skin, rarely burns, tans darkly easily; skin phototype VI = dark brown or black skin, never burns, always tans darkly.
  Participants
    Phototype I | 3
    Phototype II | 32
    Phototype III | 23
    Phototype IV | 9
Acne Duration [Mean (Standard Deviation); unit: years] | 6.8 (4.2)

OUTCOME MEASURES:

1. Primary Outcome: Part 1: Total Atrophic Acne Scar Count Per Half-face
Description: The scars were counted according to their size defined in two categories using 2-millimeter (mm) and 4-mm punch biopsy tools for size classification: 1) atrophic scars 2 to 4 mm: included boxcar (sheer edges), rolling (irregular surface), and undetermined types; 2) atrophic scars greater than (>) 4 mm: included boxcar (sheer edges), rolling (irregular surface), and undetermined types. Each type of atrophic acne scar was counted separately for each half-face by the evaluator for following regions: right forehead, right cheek, right side of the chin, left forehead, left cheek and left side of the chin. To obtain the total number of atrophic scars per half-face, atrophic acne scar counts for each half-face was added.
Time Frame: Week 24
Population: The Intent-to-Treat efficacy population (ITT) included entire population enrolled and randomized.
Measure: Mean (Standard Deviation); unit: atrophic acne scars
Groups:
- Part 1: ABPO Forte Gel: Participants applied once-daily ABPO Forte gel on half-face based on randomization (right or left side of the face) at night for 24 weeks.
- Part 1: ABPO Forte Vehicle Gel: Participants applied once-daily ABPO Forte vehicle gel on half-face based on randomization (right or left side of the face) at night for 24 weeks.
Arm/Group | Part 1: ABPO Forte Gel | Part 1: ABPO Forte Vehicle Gel
Number analyzed (Participants) | 67 | 67
atrophic acne scars | 9.5 (5.5) | 13.3 (7.4)
Statistical Analysis 1: Comparison: Part 1: ABPO Forte Gel vs Part 1: ABPO Forte Vehicle Gel; Test type: Superiority; p < 0.0001, Wilcoxon (Mann-Whitney)

2. Secondary Outcome: Part 1 and Part 2: Total Atrophic Acne Scar Count Per Half-face at Each Post-baseline Visit
Description: The scars were counted according to their size defined in two categories using 2 mm and 4 mm punch biopsy tools for size classification: 1) atrophic scars 2 to 4 mm: included boxcar (sheer edges), rolling (irregular surface), and undetermined types; 2) atrophic scars > 4 mm: included boxcar (sheer edges), rolling (irregular surface), and undetermined types. Each type of atrophic acne scar was counted separately for each half-face by the evaluator for following regions: right forehead, right cheek, right side of the chin, left forehead, left cheek and left side of the chin. To obtain the total number of atrophic scars per half-face, atrophic acne scar counts for each half-face was added.
Time Frame: Part 1: Weeks 1, 4, 8, 12, 16 and 20; Part 2: Weeks 1, 4, 8, 12, 16, 20, 36 and 48
Population: ITT population included entire population enrolled and randomized. Here, "Number Analyzed" signifies those participants who were evaluable for this outcome measure at specified time points.
Measure: Mean (Standard Deviation); unit: atrophic acne scars
Groups:
- Part 2: ABPO Forte Gel: Participants applied once-daily ABPO Forte gel on whole face for 48 weeks.
- Part 2: ABPO Forte Vehicle Gel: Participants applied once-daily ABPO Forte vehicle gel on whole face for 48 weeks.
Arm/Group | Part 1: ABPO Forte Gel | Part 1: ABPO Forte Vehicle Gel | Part 2: ABPO Forte Gel | Part 2: ABPO Forte Vehicle Gel
Number analyzed (Participants) | 67 | 67 | 45 | 45
atrophic acne scars
  Week 1 | 11.7 (6.5) | 12.8 (6.8) | 12.2 (6.6) | 13.1 (6.5)
  Week 4 | 11.9 (6.8) | 13.6 (8.0) | 12.2 (6.8) | 14.2 (8.1)
  Week 8 | 11.3 (6.7) | 13.5 (7.6) | 11.8 (7.3) | 14.0 (7.8)
  Week 12 | 10.7 (6.1) | 13.8 (7.7) | 11.3 (6.8) | 14.4 (8.1)
  Week 16 | 10.7 (6.2) | 13.7 (7.2) | 11.0 (6.8) | 14.2 (7.6)
  Week 20 | 10.3 (5.9) | 13.4 (7.5) | 10.4 (6.5) | 13.9 (8.1)
  Week 36: number analyzed (Participants) | 0 | 0 | 45 | 45
  Week 36 |  |  | 8.8 (5.3) | 11.7 (7.0)
  Week 48: number analyzed (Participants) | 0 | 0 | 45 | 45
  Week 48 |  |  | 8.4 (5.4) | 9.9 (6.3)

3. Secondary Outcome: Part 1 and Part 2: Percent Change From Baseline in Total Atrophic Acne Scar Count Per Half-face at Each Post-baseline Visit
Description: The scars were counted according to their size defined in two categories using 2 mm and 4 mm punch biopsy tools for size classification: 1) atrophic scars 2 to 4 mm: included boxcar (sheer edges), rolling (irregular surface), and undetermined types; 2) atrophic scars > 4 mm: included boxcar (sheer edges), rolling (irregular surface), and undetermined types. Each type of atrophic acne scar was counted separately for each half-face by the evaluator for following regions: right forehead, right cheek, right side of the chin, left forehead, left cheek and left side of the chin.
Time Frame: Part 1: Weeks 1, 4, 8, 12, 16, 20 and 24; Part 2: Weeks 1, 4, 8, 12, 16, 20, 24, 36 and 48
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Part 1: ABPO Forte Gel | Part 1: ABPO Forte Vehicle Gel | Part 2: ABPO Forte Gel | Part 2: ABPO Forte Vehicle Gel
Number analyzed (Participants) | 67 | 67 | 45 | 45
percent change
  Week 1 | -2.5 (12.5) | 5.8 (19.5) | -2.6 (14.2) | 6.6 (22.3)
  Week 4 | -1.0 (21.9) | 9.8 (28.1) | -0.3 (25.6) | 12.5 (31.1)
  Week 8 | -4.5 (27.4) | 12.3 (32.5) | -3.6 (32.0) | 13.0 (35.8)
  Week 12 | -7.3 (32.9) | 16.2 (40.7) | -7.1 (37.3) | 18.1 (46.4)
  Week 16 | -7.0 (35.9) | 17.1 (45.6) | -8.4 (40.7) | 18.3 (52.2)
  Week 20 | -8.7 (39.2) | 15.2 (51.7) | -11.7 (44.9) | 14.6 (58.5)
  Week 24 | -15.5 (38.9) | 14.4 (53.0) | -21.7 (42.8) | 16.7 (62.7)
  Week 36: number analyzed (Participants) | 0 | 0 | 45 | 45
  Week 36 |  |  | -25.0 (37.1) | -1.8 (52.4)
  Week 48: number analyzed (Participants) | 0 | 0 | 45 | 45
  Week 48 |  |  | -26.9 (39.7) | -15.2 (49.6)

4. Secondary Outcome: Part 1 and Part 2: Investigator's Scar Global Assessment (ISGA) Score
Description: ISGA was an assessment scale used to evaluate facial acne severity. ISGA was recorded using a 5-point scale ranges from 0 to 4, where (0 = clear [No visible scars from acne); 1 = almost clear [Hardly visible scars from 50 cm away]; 2 = mild [Easily recognizable; less than half the affected face area]; 3 = moderate [More than half and less than 75% of the affected face area]; 4 = severe [More than 75% of the affected face area]) based on inflammation, pustules and papulation/infiltration. Higher score indicated severe acne.
Time Frame: Part 1: Weeks 1, 4, 8, 12, 16, 20 and 24; Part 2: Weeks 1, 4, 8, 12, 16, 20, 24, 36 and 48
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Arm/Group | Part 1: ABPO Forte Gel | Part 1: ABPO Forte Vehicle Gel | Part 2: ABPO Forte Gel | Part 2: ABPO Forte Vehicle Gel
Number analyzed (Participants) | 67 | 67 | 45 | 45
score on a scale
  Week 1 | 2.3 (0.6) | 2.3 (0.6) | 2.3 (0.7) | 2.3 (0.7)
  Week 4 | 2.2 (0.6) | 2.3 (0.7) | 2.2 (0.7) | 2.2 (0.8)
  Week 8 | 2.2 (0.6) | 2.3 (0.7) | 2.2 (0.7) | 2.3 (0.7)
  Week 12 | 2.0 (0.7) | 2.2 (0.6) | 1.9 (0.7) | 2.2 (0.6)
  Week 16 | 2.0 (0.7) | 2.2 (0.6) | 1.9 (0.7) | 2.1 (0.6)
  Week 20 | 1.9 (0.7) | 2.1 (0.7) | 1.8 (0.8) | 2.0 (0.8)
  Week 24 | 1.8 (0.8) | 2.1 (0.7) | 1.6 (0.8) | 2.0 (0.8)
  Week 36: number analyzed (Participants) | 0 | 0 | 45 | 45
  Week 36 |  |  | 1.5 (0.7) | 1.8 (0.6)
  Week 48: number analyzed (Participants) | 0 | 0 | 45 | 45
  Week 48 |  |  | 1.4 (0.8) | 1.5 (0.7)

5. Secondary Outcome: Part 1: Percentage of Participants With Investigator's Preference on Overall Scar Severity
Description: The investigator rated their preference on a scale ranging from -2 (left side a lot better than right) to 2 (right side a lot better than left). Overall scar severity was assessed using a 5-point scale where (-2 = Left a lot better than right; -1 = Left a little bit better than right; 0 = No preference; 1 = Right a little bit better than left; 2 = Right a lot better than left. ABPO forte was applied on left side and vehicle gel was applied on right side.
Time Frame: At Week 12 and Week 24
Population: ITT population included entire population enrolled and randomized. Here, "Overall Number of Participants Analyzed" signifies those participants who were evaluable for this outcome measure and "Number analyzed" signifies those participants who were evaluable for this outcome measure at the specified time point.
Measure: Number; unit: percentage of participants
Groups:
- Part 1: All Participants: Participants applied once-daily ABPO Forte gel on half-face and ABPO Forte vehicle gel on the other side of the face based on randomization (right or left side of the face) at night for 24 weeks.
Arm/Group | Part 1: All Participants
Number analyzed (Participants) | 63
percentage of participants
  Week 12: ABPO Forte a lot better than Vehicle: number analyzed (Participants) | 59
  Week 12: ABPO Forte a lot better than Vehicle | 5.1
  Week 12: ABPO Forte a little bit better than Vehicle: number analyzed (Participants) | 59
  Week 12: ABPO Forte a little bit better than Vehicle | 33.9
  Week 24: ABPO Forte a lot better than Vehicle | 17.5
  Week 24: ABPO Forte a little bit better than Vehicle | 36.5

6. Secondary Outcome: Part 1 and Part 2: Percent Change From Baseline in Total Lesion Count Per Half-face at Each Post-baseline Visit
Description: Total lesion counts corresponded to the sum of inflammatory and non-inflammatory lesions, and other lesions. The investigator counted all inflammatory lesions (papules and pustules), non-inflammatory lesions (open and closed comedone) and other lesions (nodules) for each half-face.
Time Frame: Part 1: Weeks 1, 4, 8, 12, 16 and 20; Part 2: Weeks 1, 4, 8, 12, 16, 20, 36 and 48
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Part 1: ABPO Forte Gel | Part 1: ABPO Forte Vehicle Gel | Part 2: ABPO Forte Gel | Part 2: ABPO Forte Vehicle Gel
Number analyzed (Participants) | 67 | 67 | 45 | 45
percent change
  Week 1 | -20.9 (22.1) | -5.7 (19.9) | -23.4 (22.4) | -7.6 (19.7)
  Week 4 | -34.1 (27.4) | -13.1 (29.1) | -38.6 (24.4) | -15.2 (29.3)
  Week 8 | -45.7 (29.3) | -25.3 (31.4) | -53.6 (23.2) | -30.4 (28.9)
  Week 12 | -54.5 (27.9) | -32.9 (32.7) | -63.3 (21.6) | -38.7 (31.7)
  Week 16 | -60.4 (28.5) | -35.4 (35.9) | -71.9 (19.2) | -43.3 (36.2)
  Week 20 | -63.7 (28.0) | -43.2 (33.5) | -75.0 (16.4) | -53.2 (29.0)
  Week 24 | -66.7 (29.1) | -45.8 (33.6) | -79.4 (16.1) | -56.4 (29.4)
  Week 36: number analyzed (Participants) | 0 | 0 | 45 | 45
  Week 36 |  |  | -74.0 (19.2) | -69.9 (23.8)
  Week 48: number analyzed (Participants) | 0 | 0 | 45 | 45
  Week 48 |  |  | -72.7 (22.8) | -70.4 (23.1)

7. Secondary Outcome: Part 1 and Part 2: Percent Change From Baseline in Inflammatory Lesion Count Per Half-face at Each Post-baseline Visit
Description: Inflammatory lesions included papules and pustules. Papule is a small, solid elevation less than one centimeter in diameter. Most of the lesion is above the surface of the skin. Pustule is a small, circumscribed elevation of the skin which contains yellow-white exudates.
Time Frame: Part 1: Weeks 1, 4, 8, 12, 16, 20 and 24; Part 2: Weeks 1, 4, 8, 12, 16, 20, 24, 36 and 48
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Part 1: ABPO Forte Gel | Part 1: ABPO Forte Vehicle Gel | Part 2: ABPO Forte Gel | Part 2: ABPO Forte Vehicle Gel
Number analyzed (Participants) | 67 | 67 | 45 | 45
percent change
  Week 1 | -28.0 (33.0) | -10.4 (24.8) | -29.2 (34.4) | -11.9 (26.7)
  Week 4 | -43.5 (30.8) | -19.8 (36.7) | -50.1 (24.4) | -19.6 (39.2)
  Week 8 | -55.1 (35.0) | -31.2 (34.7) | -67.9 (17.4) | -36.7 (32.5)
  Week 12 | -63.6 (33.0) | -39.1 (37.9) | -74.9 (21.2) | -47.8 (32.4)
  Week 16 | -70.1 (29.6) | -39.4 (39.6) | -82.6 (14.6) | -51.3 (35.6)
  Week 20 | -72.6 (30.7) | -47.5 (37.5) | -84.6 (17.4) | -60.2 (27.5)
  Week 24 | -75.4 (29.8) | -50.2 (36.3) | -88.5 (11.1) | -64.0 (23.2)
  Week 36: number analyzed (Participants) | 0 | 0 | 45 | 45
  Week 36 |  |  | -81.3 (20.5) | -75.5 (25.5)
  Week 48: number analyzed (Participants) | 0 | 0 | 45 | 45
  Week 48 |  |  | -77.2 (27.1) | -73.3 (25.7)

8. Secondary Outcome: Part 1 and Part 2: Percent Change From Baseline in Non-inflammatory Lesion Count Per Half-face at Each Post-baseline Visit
Description: Non-inflammatory lesions included open comedone and closed comedone. Open comedone is a mass of sebaceous material that is impacted behind an open follicular orifice (blackhead). Closed comedone is a mass of sebaceous material that is impacted behind a closed follicular orifice (white head).
Time Frame: Part 1: Weeks 1, 4, 8, 12, 16, 20 and 24; Part 2: Weeks 1, 4, 8, 12, 16, 20, 24, 36 and 48
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: percent change
Arm/Group | Part 1: ABPO Forte Gel | Part 1: ABPO Forte Vehicle Gel | Part 2: ABPO Forte Gel | Part 2: ABPO Forte Vehicle Gel
Number analyzed (Participants) | 67 | 67 | 45 | 45
percent change
  Week 1: number analyzed (Participants) | 66 | 67 | 45 | 45
  Week 1 | -9.2 (29.2) | 0.3 (30.8) | -10.7 (33.1) | -2.7 (33.6)
  Week 4 | -20.1 (36.1) | -1.5 (36.8) | -22.8 (39.4) | -4.7 (39.1)
  Week 8 | -32.4 (34.7) | -16.0 (42.7) | -36.5 (36.4) | -21.7 (44.8)
  Week 12 | -40.8 (31.3) | -21.1 (37.9) | -47.8 (29.9) | -24.4 (40.7)
  Week 16 | -47.7 (34.1) | -24.7 (40.8) | -58.9 (30.1) | -29.7 (43.8)
  Week 20 | -51.4 (33.1) | -33.3 (39.9) | -62.4 (27.6) | -41.7 (39.9)
  Week 24 | -55.4 (34.7) | -35.6 (40.5) | -67.9 (28.2) | -44.6 (41.0)
  Week 36: number analyzed (Participants) | 0 | 0 | 45 | 45
  Week 36 |  |  | -64.5 (28.6) | -59.6 (30.8)
  Week 48: number analyzed (Participants) | 0 | 0 | 45 | 45
  Week 48 |  |  | -64.9 (27.6) | -62.5 (28.4)

9. Secondary Outcome: Part 1 and Part 2: Investigator's Global Assessment (IGA) Score Per Half-face at Each Post-baseline Visit
Description: IGA is an assessment scale used to determine severity of acne and clinical response to treatment on a 5-point scale (0 = clear [Clear skin with no inflammatory or non inflammatory lesions]; 1= almost clear [A few scattered comedones and a few small papules]; 2= mild [Easily recognizable; less than half the face is involved. Some comedones and some papules and pustules]; 3= moderate [More than half of the face is involved. Many comedones, papules and pustules. One small nodule may be present] and 4= severe [Entire face is involved. Covered with comedones, numerous papules and pustules. Few nodules may or may not be present]) based on erythema and papulation/ infiltration. Therapeutic response is an IGA score of 0 (clear) or 1 (almost clear).
Time Frame: Part 1: Weeks 1, 4, 8, 12, 16, 20 and 24; Part 2: Weeks 1, 4, 8, 12, 16, 20, 24, 36 and 48
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: score on a scale
Groups:
- Part 1: A BPO Forte Gel: Participants applied once-daily ABPO Forte gel on half-face based on randomization (right or left side of the face) at night for 24 weeks.
Arm/Group | Part 1: A BPO Forte Gel | Part 1: ABPO Forte Vehicle Gel | Part 2: ABPO Forte Gel | Part 2: ABPO Forte Vehicle Gel
Number analyzed (Participants) | 67 | 67 | 45 | 45
score on a scale
  Week 1 | 2.7 (0.6) | 3.0 (0.4) | 2.7 (0.6) | 3.0 (0.4)
  Week 4 | 2.5 (0.7) | 2.8 (0.6) | 2.5 (0.7) | 2.8 (0.6)
  Week 8 | 2.3 (0.7) | 2.7 (0.6) | 2.1 (0.8) | 2.6 (0.6)
  Week 12 | 1.9 (0.8) | 2.4 (0.7) | 1.7 (0.7) | 2.2 (0.7)
  Week 16 | 1.6 (0.8) | 2.2 (0.8) | 1.2 (0.5) | 2.0 (0.9)
  Week 20 | 1.5 (0.9) | 2.1 (0.8) | 1.1 (0.6) | 1.9 (0.8)
  Week 24 | 1.4 (0.9) | 2.2 (0.8) | 1.0 (0.5) | 1.9 (0.8)
  Week 36: number analyzed (Participants) | 0 | 0 | 45 | 45
  Week 36 |  |  | 1.2 (0.6) | 1.4 (0.7)
  Week 48: number analyzed (Participants) | 0 | 0 | 45 | 45
  Week 48 |  |  | 1.2 (0.7) | 1.3 (0.7)

ADVERSE EVENTS:
Time Frame: Part 1: up to 24 weeks; Part 2: up to 48 weeks
Description: The safety population included all randomized participants, after exclusion of participants who never took the treatment with certainty based on monitoring report.
Arm/Group | Part 1: ABPO Forte Gel | Part 1: ABPO Forte Vehicle Gel | Part 2: ABPO Forte Gel | Part 2: ABPO Forte Vehicle Gel
All-Cause Mortality (participants affected / at risk) | 0/67 | 0/67 | 0/45 | 0/45
Serious Adverse Events (participants affected / at risk) | 0/67 | 0/67 | 0/45 | 0/45
Other Adverse Events (participants affected / at risk) | 11/67 | 5/67 | 14/45 | 0/45
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Part 1: ABPO Forte Gel (N=67) | Part 1: ABPO Forte Vehicle Gel (N=67) | Part 2: ABPO Forte Gel (N=45) | Part 2: ABPO Forte Vehicle Gel (N=45)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 6 | 0
Headache (Nervous system disorders) | 0 (0) | 0 (0) | 5 | 0
Skin irritation (Skin and subcutaneous tissue disorders) | 11 (11) | 5 (5) | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other

DOCUMENTS (2):
  • Study Protocol (2016-07-06): https://cdn.clinicaltrials.gov/large-docs/21/NCT02735421/Prot_000.pdf
  • Statistical Analysis Plan (2017-06-27): https://cdn.clinicaltrials.gov/large-docs/21/NCT02735421/SAP_001.pdf